CLINICAL TRIAL: NCT05559125
Title: An Open-label, Single-ascending Dose Phase I Study to Evaluate the Safety and Tolerability of STSA-1002 Combined With STSA-1005 in Healthy Subjects
Brief Title: A Study of STSA-1002 Combined With STSA-1005 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the COVID-19 epidemic situation, the sponsor has decided to terminate the project.
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1002/1005-01
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-12

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- STSA-1002 and STSA-1005 dose level 1 (Experimental)
  Interventions: Drug: STSA-1002 Injection; Drug: STSA-1005 Injection
- STSA-1002 and STSA-1005 dose level 2 (Experimental)
  Interventions: Drug: STSA-1002 Injection; Drug: STSA-1005 Injection
- STSA-1002 and STSA-1005 dose level 3 (Experimental)
  Interventions: Drug: STSA-1002 Injection; Drug: STSA-1005 Injection
- STSA-1002 and STSA-1005 dose level 4 (Experimental)
  Interventions: Drug: STSA-1002 Injection; Drug: STSA-1005 Injection

INTERVENTIONS:
Drug: STSA-1002 Injection — Intravenous injection
Drug: STSA-1005 Injection — Intravenous injection

SUMMARY:
An open-label, single-ascending dose phase I study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of STSA-1002 combined with STSA-1005 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, aged ≥ 18 but ≤ 45, male and female;
* Weight: Male≥50.0kg, Female ≥ 45kg; Body mass index: 19.0-26.0 kg/m2, inclusive;
* Subjects (including their partners) must take effective contraceptive measures and have no birth plan or sperm or egg donation plan during the trial period and within 6 months after the end of the last administration;
* The subjects were aware of the risks of the trial, voluntarily participated in the study and signed the informed consent form (ICF).

Exclusion Criteria:

* Have a history of serious disease (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular diseases) or have undergone any major surgery within 2 months prior to screening;
* The investigators determined that abnormalities in pre-enrollment physical examinations, laboratory tests, and trial-related tests were clinically significant;
* A definite history of food or drug allergies;
* Positive screening test results for human immunodeficiency virus (HIV) antibodies, syphilis-specific antibody, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb);
* History of tuberculosis; or combined with T-SPOT.TB results, low-dose chest CT comprehensive evaluation of tuberculosis infection;
* Hemoglobin was lower than the lower limit of normal value during the screening period;
* Smoking more than 5 or equivalent cigarettes per day in the 3 months before screening;
* Regular drinkers in the 6 months prior to screening, i.e. those who have consumed more than 2 units of alcohol per day (1 unit =360ml beer or 45ml spirits with an alcohol concentration of 40% or 150ml wine) in the 6 months prior to screening or have a positive alcohol test result;
* Subjects with a history of substance abuse within 1 year before screening or have a positive drug test result;
* Blood loss or blood donation > 400ml three months before screening, or blood transfusion history within 4 weeks before inclusion;
* Participate in clinical trials of new drugs or vaccines as a subject within 3 months prior to screening；
* Vaccination was given within 1 month before screening or planned between the study period and 2 months after the end of the study;
* Use of medications that may affect immune function in the 6 months prior to screening or any monoclonal antibody or biologic treatment in the 3 months prior to screening and use of prescription drugs/over-the-counter drugs or herbal medicines in the 14 days prior to screening；
* Drink more than 5 cups of coffee, tea or cola (150ml or more per cup) daily within 3 months before screening;
* Pregnant or lactating women;
* A history of blood and needle sickness；
* Other circumstances in which the investigator considers it inappropriate to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram、Vital Signs And Physical Examination Abnormalities. | 56 days
  To evaluate the safety and tolerability of single intravenous administration of STSA-1002 combined with STSA-1005 in healthy adult subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax). | Up to 1344hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Time of maximum concentration (Tmax) | Up to 1344hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Elimination half-life (t1/2). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Elimination rate constant (Kel). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Clearance (CL). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Apparent volume of distribution (Vz). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Mean residence time (MRTlast). | Up to 1344 hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Extrapolated area under the curve (AUC_%Extrap). | Up to 1344hours postdose
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 combined with STSA-1005 in healthy adult subjects.
Change from baseline in concentration of free C5a and anti-drug antibody. | Up to 1344 hours postdose
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 combined with STSA-1005 in healthy subjects.
Change from baseline in concentration of cytokine (IL-2, IL-6, IL-8, IL-10, TNF-α, IFN-γ, GM-CSF). | Up to 1344 hours postdose
  To evaluate the effects of STSA-1002 combined with STSA-1005 on cytokine (IL-2, IL-6, IL-8, IL-10, TNF-α, IFN-γ, GM-CSF).

CONTACTS AND LOCATIONS:
Overall Officials: Fengxue Guo, Bachelor, Principal Investigator — The Second Affiliated Hospital of Xingtai Medical College
Locations (1):
- The Second Affiliated Hospital Of Xingtai Medical College, Xingtai, Hebei, China